CLINICAL TRIAL: NCT02302768
Title: Effect of Supplementation of Two Doses of L-selenomethionine (Semet; 80 and 160 mcg) Versus Placebo in Patients With Chronic Autoimmune Thyroiditis (AIT) With Normal Thyroid Function.
Brief Title: Effect of Semet (80 and 160 mcg) Versus Placebo in Euthyroid Patients With AIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Collaborators: IBSA Institut Biochimique SA (Industry)
Responsible Party: Principal Investigator, Furio Pacini, Full Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SELENIO 2012
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Thyroiditis Autoimmune
MeSH Terms: conditions — Hashimoto Disease | interventions — Selenomethionine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Patients randomized to receive same pharmaceutical form (capsule) used for the two Semet groups, with the same excipients but the active drug.
  Interventions: Other: Placebo
- 80-Semet (Active Comparator): Patients randomized to receive selenomethionine at 80 mcg per day.
  Interventions: Dietary Supplement: Selenomethionine
- 160-Semet (Active Comparator): Patients randomized to receive selenomethionine at 160 mcg per day.
  Interventions: Dietary Supplement: Selenomethionine

INTERVENTIONS:
Dietary Supplement: Selenomethionine
  Arms: 160-Semet; 80-Semet
Other: Placebo
  Arms: Placebo

SUMMARY:
Over the past 10 years, several clinical studies have suggested that selenium supplementation may influence the natural history of AIT. Recently, Interferon gamma (IFNγ)-inducible chemokines (CXCL-9, -10 and -11) were shown to be elevated in the AIT patients. The aim of this prospective, randomized, controlled study is to evaluate the effect of two different doses of selenomethionine (80 or 160 mcg) versus placebo in euthyroid women with AIT, in terms of reduction of anti-thyroid antibodies and improvement of thyroid hypoechogenicity, over 24 months. Serum levels of selenium, CXCL-9, -10 and -11 and their regulators, Tumor necrosis factor alpha (TNFα) and INFγ, thyroid function and volume and the quality of life of AIT patients are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic autoimmune thyroiditis defined by positivity of anti thyroperoxidase and/or anti thyroglobulin antibodies (> or = 100 U/l) and thyroid hypoechogenicity

Exclusion Criteria:

* Presence of other thyroid disease but micronodules
* History of the malignancy in the past 5 years
* Drugs affecting immune system and/or thyroid function
* Pregnancy detected during screening or follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of anti-thyroid antibodies | 12 months
  Anti thyroperoxidase and thyroglobulin antibodies are measured by a chemiluminescent assay. Any statistically significant decrease of one or both antibody values compared to the baseline is considered a reduction relevant to the study outcome.
Improvement of thyroid echogenicity | 12 months
  High-resolution sonograhic images are captured, converted into a spectrum of gray-scale pixels (gsp) ranging from 0 (lowest echogenicity) to 255 (highest echogenicity) and a mean value is then obtained. Any statistically significant increase of the gsp compared to the baseline is considered an improvement relevant to the study outcome.

SECONDARY OUTCOMES:
Prevention or reduction of the incidence of hypothyroidism | 24 months
  Defined by a significant lower number of new subclinical or overt hypothyroidism cases in the two Semet groups compared to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Furio Pacini, MD, Principal Investigator — University of Siena

REFERENCES:
- [Background] Rayman MP. Selenium and human health. Lancet. 2012 Mar 31;379(9822):1256-68. doi: 10.1016/S0140-6736(11)61452-9. Epub 2012 Feb 29. PMID 22381456
- [Background] Nacamulli D, Petricca D, Mian C. Selenium and autoimmune thyroiditis. J Endocrinol Invest. 2013 Nov;36(10 Suppl):8-14. PMID 24419054
- [Background] Rotondi M, Chiovato L. The chemokine system as a therapeutic target in autoimmune thyroid diseases: a focus on the interferon-gamma inducible chemokines and their receptor. Curr Pharm Des. 2011;17(29):3202-16. doi: 10.2174/138161211798157559. PMID 21864266